CLINICAL TRIAL: NCT02331147
Title: A Prospective, Randomized, Comparative Parallel Study of Allogenic Dermis Graft in the Management of Diabetic Foot Ulcers
Brief Title: Allogenic Dermis Versus Standard Care in the Management of Diabetic Foot Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Musculoskeletal Transplant Foundation (Other)
Collaborators: Professional Education and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20142081
Record Dates: First submitted 2014-12-29; First posted 2015-01-06 (Estimated); Last update posted 2022-06-01 (Actual); Status verified 2018-01

CONDITIONS: Diabetic; Foot Ulcers
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of Care (Sham Comparator): Surgical debridement of DFU, The wound will be debrided and cleaned. Patient ulcers will be assessed and measured weekly in cm length by width. Application of collagen alginate and gauze dressing application to be changed daily by patient. Patient will practice off loading
  Interventions: Other: Offloading
- Human Dermis (Active Comparator): Application of Human Allogenic Dermis with Dressing Application, to be changed weekly. Patient would will be measured in cm length by width weekly Patient will practice Offloading.
  If the ulcer has not closed completely, an additional piece of Human Dermis will be applied weekly at weeks 2-11 in a similar fashion
  Interventions: Other: Offloading; Other: Dressing Application

INTERVENTIONS:
Other: Offloading — Patient will be offloaded in a diabetic camboot after treatment
Other: Dressing Application — Application of a non-adherent dressing, a moisture retentive dressing, and a multi-layer compression dressing.
  Arms: Human Dermis

SUMMARY:
This is comparison trial comparing human dermis to standard wound care for non healing diabetic wound

DETAILED DESCRIPTION:
This is a prospective, randomized, comparative, parallel group, Multi-center clinical trial comparing the proportion of ulcers completely healed by use of allogenic dermal graft versus the standard protocol of wound care in diabetic patients with a diabetic foot ulcer with adequate arterial perfusion, for wound healing to the affected limb. The primary objective of this study is to compare the proportion of ulcers completely healed by the allogenic dermal graft protocol of care to the standard protocol of care in the management of indolent diabetic ulcers at 6 weeks. The secondary objectives of this study are to compare the proportion of healing at 4 weeks, 12 weeks and, the mean time to healing. Patient after signing IRB approve informed consent, upon meeting inclusion/exclusion criteria will be randomized into one of two group. One group receiving standard of care protocol, with an offloading boot, and one group received human allogenic dermis application, with compressive dressing and offloading boot. Patients will be seen weekly or until complete healing occurs. Measurements will be taken of the diabetic ulcers using the a centimeter ruler measuring length by width.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age 18 or older.
2. Patient is willing to provide informed consent and is willing to participate in all procedures and follow up evaluations necessary to complete the study.
3. Patient's ulcer must be diabetic in origin and larger than 1 cm2.
4. Patients with Type 1 or Type 2 diabetes (criteria for the diagnosis of diabetes mellitus per ADA).
5. Ulcer must be present for a minimum of four weeks before enrollment randomization, with documented failure of conventional ulcer therapy to heal the wound.
6. A two week run-in period will precede enrollment/ randomization in the trial to document the indolent nature of the wounds selected.
7. Additional wounds may be present but not within 3 cm of the study wound.
8. Wound must be present anatomically on the foot as defined by beginning below the malleoli of the ankle and be neuropathic in origin.
9. Patient's ulcer must exhibit no clinical signs of infection.
10. Serum Creatinine less than 3.0mg/dl within last six months.
11. HbA1c less than or equal to 12% within last 90 days.
12. Patient has adequate circulation to the affected extremity, as demonstrated by one of the following within the past 60 days:

    1. Dorsum transcutaneous oxygen test (TcPO2) with results ≥30mmHg,
    2. ABIs with results of ≥0.7 and ≤1.2, OR
    3. Doppler arterial waveforms, which are triphasic or biphasic at the ankle of affected leg.

Exclusion Criteria:

1. Patients presenting with an ulcer probing to tendon, muscle, capsule or bone (UT Grade IIIA-D). A positive probe-to-bone will be confirmed when bone or joint can be felt with a sterile, ophthalmological probe.
2. Patients whose index diabetic foot ulcers are greater than 25 cm2.
3. Patients considered not in reasonable metabolic control, confirmed by an HbA1c greater than 12% within previous 90 days.
4. Patients whose serum creatinine levels are 3.0mg/dl or greater within the last six months.
5. Patients with a known history of poor compliance with medical treatments.
6. Patients who have been previously randomized into this study, or are presently participating in another clinical trial.
7. Patients who are currently receiving radiation therapy or chemotherapy.
8. Patients with known or suspected local skin malignancy to the index diabetic ulcer.
9. Patients diagnosed with autoimmune connective tissues diseases.
10. Non-revascularizable surgical sites.
11. Active infection at site.
12. Any pathology that would limit the blood supply and compromise healing.
13. Patients that have received a biomedical or topical growth factor for their wound within the previous 30 days.
14. Patients who are pregnant or breast feeding.
15. Patients who are taking medications that are considered immune system modulators which could affect graft incorporation.
16. Patients with known hypersensitivity to components of any treatment used in the trial.
17. Wounds greater than one year in duration without intermittent healing.
18. Wounds improving greater than 20% over the first two weeks (run-in period) of the trial using standard of care dressing and camboot.
19. Patients taking Cox-2 inhibitors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
proportion of ulcers completely healed by the allogenic dermal graft protocol of care to the standard protocol of care in the management of indolent diabetic ulcers at 6 weeks | 6 weeks

SECONDARY OUTCOMES:
Compare the proportion of ulcers completely healed at 4 weeks | 4 weeks
Compare the proportion of ulcers completely healed at 12 weeks | 12 weeks
Mean time to healing | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Charles M Zelen, DPM, Principal Investigator — CEO; Professional Education and Research Institute
Locations (3):
- United States (3):
  - Shenandoah Lower Extremity Research, Roanoke, Virginia
  - Professional Education and Research Institute, Roanoke, Virginia
  - Foot and Ankle Associates of Southwest VA, Salem, Virginia